CLINICAL TRIAL: NCT03714815
Title: A Long-term, Multicenter, Single-arm, Open-label Extension of the SERENADE Study, to Assess the Safety and Efficacy of Macitentan in Subjects With Heart Failure With Preserved Ejection Fraction and Pulmonary Vascular Disease
Brief Title: A Long Term Study to Find Out if Macitentan is an Effective and Safe Treatment for Patients With Heart Failure With Preserved Ejection Fraction and Pulmonary Vascular Disease
Acronym: SERENADE OL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: the absence of a positive trend in all efficacy parameters indicates that macitentan 10 mg does not have a beneficial effect in patients with HFpEF and PVD.
Sponsor: Actelion (Industry)
Collaborators: Almac Clinical Technologies (Industry); Frontier Science & Technology Research Foundation, Inc. (Industry); Covance (Industry); Chiltern International Ltd. (Industry); WorldCare Clinical, LLC (Industry); AcitGraph (Other); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055G203; 2018-001603-37 (EudraCT Number)
Record Dates: First submitted 2018-10-19; First posted 2018-10-22 (Actual); Results first posted 2022-11-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction and Pulmonary Vascular Disease
Keywords: pulmonary vascular disease; macitentan; heart failure with preserved ejection fraction
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Intervention Model Description: Subjects who remained in main study (SERENADE/AC-055G202, NCT03153111) after randomization and who meet the eligibility criteria described will be eligible to enter this single-arm OL extension study. All enrolled subjects will receive macitentan 10 mg. For this OL extension study no primary efficacy endpoint has been defined and all efficacy endpoints are of exploratory nature. The ones listed below are considered safety endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-label treatment period (Experimental): oral administration of 10 mg macitentan once daily
  Interventions: Drug: macitentan 10 mg

INTERVENTIONS:
Drug: macitentan 10 mg — macitentan 10 mg, film-coated tablet, oral use

SUMMARY:
The aim of this open-label (OL) extension trial is to study the long-term safety and efficacy of macitentan in subjects with heart failure with preserved ejection fraction (HFpEF) and pulmonary vascular disease (PVD) beyond the treatment in the double-blind parent SERENADE study (AC-055G202, NCT03153111). Furthermore, this OL extension study will give eligible subjects of the main study (SERENADE/AC-055G202, NCT03153111) an opportunity to continue or start receiving macitentan.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Informed Consent Form (ICF).
* Participant remained in the main study (SERENADE/AC-055G202, NCT03153111) for: a) 52 weeks after randomization if entered this Open-label (OL) extension study prior to protocol Version 4, b) At least 24 weeks after randomization if entering this OL extension study under protocol Version 4
* A woman of childbearing potential is eligible only if: (1) Negative pre-treatment serum pregnancy test; (2) Agreement to undertake monthly pregnancy tests from the enrollment visit up to at least 30 days after study treatment discontinuation; and (2) Agreement to use reliable contraception from at least 30 days prior to the enrollment visit up to at least 30 days after study treatment discontinuation.

Exclusion Criteria:

* Premature discontinuation of study treatment in the main study (SERENADE/AC-055G202, NCT03153111) due to an adverse event related to: (1) Edema or fluid retention; (2) Worsening of heart failure; (3) Liver aminotransferase elevation; and (4) Study treatment, based on investigators' discretion
* Liver aminotransferase elevations, at the enrollment visit, fulfilling the following criteria: (1) Alanine amino transferase (ALT) / aspartate aminotransferase (AST) greater than or equal to (>=) 8 * the upper limit of normal (ULN); (2) ALT/AST >= 3 * ULN and associated clinical symptoms of liver injury, for example: nausea, vomiting, fever, abdominal pain, jaundice, unusual lethargy or fatigue, flu-like syndrome (arthralgia, myalgia, fever); and (3) ALT/AST >= 3 * ULN and associated increase in total bilirubin to >= 2 * ULN
* Treatment with the following forbidden medications within 1 month prior to the enrollment visit: (1) Treatments that may interfere with the assessment of efficacy (that is, endothelin receptor antagonists, prostanoids, phosphodiesterase-5 inhibitors, guanylate cyclase stimulators); (2) Strong cytochrome P-450 3A4 (CYP3A4) inducers such as rifabutin, rifampin, rifampicin, rifapentin, carbamazepine, phenobarbital, phenytoin, or St. John's wort; (3) Strong CYP3A4 inhibitors such as ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, and saquinavir or a moderate dual CYP3A4/CYP2C9 inhibitor (for example, fluconazole or amiodarone) or co-administration of a combination of moderate CYP3A4 (for example, ciprofloxacin, cyclosporine, diltiazem, erythromycin, verapamil) and moderate CYP2C9 inhibitors (for example, miconazole, piperine), in the 1-month period prior to baseline. This will not necessarily apply to participants who are already well-managed on such an ongoing combination; and (4) any other investigational treatment
* Pregnant, planning to be become pregnant or lactating.
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results, such as drug or alcohol dependence or psychiatric disease.
* Known hypersensitivity to macitentan or drugs of the same class, or any of the study drug excipients (for example, soy lecithin, lactose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Byra, MD, Study Director — Actelion
Locations (44):
- United States (11):
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University Of Iowa - Hospitals & Clinics, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School Of Medicine, St Louis, Missouri
  - Allegheny, Pittsburgh, Pennsylvania
  - North Dallas Research Associates, McKinney, Texas
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - MultiCare Health System, Tacoma, Washington
  - Aurora Saint Lukes Medical Center, Milwaukee, Wisconsin
- Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Argentina
- Medizinische Universitaet Wien, Vienna, Austria
- Brazil (2):
  - Maestri E Kormann Consultoria Médico- Científica Ltda, Blumenau
  - Instituto do Coracao de Marília, Marília
- Bulgaria (2):
  - Diagnostic Consulting Center I Sliven, Sliven
  - Medical Centre Synexus, Sofia
- Bispebjerg Og Frederiksberg Hospital, Copenhagen, Denmark
- France (3):
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - CHU Rouen Hopital Charles Nicolle, Rouen
- Germany (3):
  - Universitätsklinikum Carl Gustav Carus Medizinische Klinik und Poliklinik 1-Pneumologie, Dresden
  - Universitaetsklinikum Giessen, Giessen
  - Universitaetsklinikum Schleswig Holstein Campus Kiel, Kiel
- Semmelweis Egyetem Varosmajor Sziv es Ergyogyaszati Klinika, Budapest, Hungary
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Poland (3):
  - Krakowski Szpital Specjalityczny im Jana Pawla II Oddzial Kliniczny Chorob Serca i Naczyn, Krakow
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego SPZOZ, Lublin
  - 4 Wojskowy Szpital Kliniczny Z Poliklinika SP ZOZ, Wroclaw
- Romania (3):
  - Cardiomed, Craiova
  - SAL MED Pitesti, Piteşti
  - Cmi Dr Podoleanu Cristian, Târgu Mureş
- Russia (4):
  - Federal State Budget Scientific Institution, Kemerovo
  - Moscow City Clinical Hospital No.51, Moscow
  - Federal State Budgetary Institution, Saint Petersburg
  - Ekaterinburg City Clinical Hospital #14, Yekaterinburg
- Sahlgrenska Universitetsjukhuset, Gothenburg, Sweden
- United Kingdom (2):
  - Royal Free Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials\transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Shah SJ, Bonderman D, Borlaug BA, Cleland JGF, Lack G, Lu W, Voors AA, Zannad F, Gladwin MT. Macitentan for Heart Failure With Preserved or Mildly Reduced Ejection Fraction and Pulmonary Vascular Disease: Results of the SERENADE Randomized Clinical Trial and Open-Label Extension Study. Circ Heart Fail. 2025 Mar;18(3):e011381. doi: 10.1161/CIRCHEARTFAILURE.123.011381. Epub 2025 Mar 11. PMID 40066571

RESULTS

PARTICIPANT FLOW:
Groups:
- Macitentan 10 mg: Eligible participants who remained in the main study (NCT03153111) for at least 24 weeks after randomization, entered this open-label extension study to receive macitentan 10 milligrams (mg) tablet orally once daily until the end of the treatment (treatment exposure ranged from 0.4 to 126 weeks).
Period: Overall Study
Arm/Group | Macitentan 10 mg
Started | 91
Completed | 76
Not Completed | 15
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — Death | 11

BASELINE CHARACTERISTICS:
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (9.21)
Age, Customized [Count of Participants; unit: Participants]
  From 18 to 64 years | 14
  From 65 to 84 years | 69
  85 years and over | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 87
  More than one race | 0
  Unknown or Not Reported | 0
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 1
  AUSTRIA | 2
  BRAZIL | 2
  BULGARIA | 8
  DENMARK | 2
  FRANCE | 5
  GERMANY | 4
  ISRAEL | 23
  POLAND | 7
  ROMANIA | 4
  RUSSIAN FEDERATION | 14
  SWEDEN | 2
  UNITED KINGDOM | 3
  UNITED STATES | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Deaths up to 30 Days After Study Treatment Discontinuation
Description: Number of participants with all-cause deaths up to 30 days after study treatment discontinuation were reported. All-cause deaths are defined as all anticipated and unanticipated deaths due to any cause.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 0.4 to 126 weeks)
Population: The safety analysis set included all participants who received at least 1 dose of macitentan 10 milligrams (mg).
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 91
Participants | 11

2. Primary Outcome: Number of Participants With All-cause Hospital Admissions up to 30 Days After Study Treatment Discontinuation
Description: Number of participants with all-cause hospital admissions up to 30 days after study treatment discontinuation were reported.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 0.4 to 126 weeks)
Population: The safety analysis set included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 91
Participants | 42

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) up to 30 Days After Study Treatment Discontinuation
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is a suspected transmission of any infectious agent via a medicinal product, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above. Any AE and SAE occurring at or after the study treatment start up to 30 days after end of treatment (EOT) within the analysis set was considered to be treatment-emergent.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 0.4 to 126 weeks)
Population: The safety analysis set included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 91
Participants
  TEAEs | 81
  TESAEs | 49

4. Primary Outcome: Number of Participants With TEAEs Leading to Premature Discontinuation of Study Treatment
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Any AE occurring at or after the study treatment start up to 30 days after EOT within the analysis set was considered to be treatment-emergent.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 0.4 to 126 weeks)
Population: The safety analysis set included all participants who received at least 1 dose of macitentan 10 mg.
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 91
Participants | 25

5. Primary Outcome: Change From Baseline in Systolic and Diastolic Arterial Blood Pressure (BP) at Week 24
Description: Change from baseline in systolic and diastolic arterial BP at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: The safety analysis set included all participants who received at least 1 dose of macitentan 10 mg. Here, "N" (number of participants analyzed) specifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 62
millimeters of mercury (mmHg)
  Systolic BP | -5.01 (13.152)
  Diastolic BP | -3.34 (9.903)

6. Primary Outcome: Change From Baseline in Systolic and Diastolic Arterial Blood Pressure (BP) at Week 52
Description: Change from baseline in systolic and diastolic arterial BP at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 53
mmHg
  Systolic BP | -2.10 (20.855)
  Diastolic BP | -0.79 (11.685)

7. Primary Outcome: Change From Baseline in Pulse Rate at Week 24
Description: Change from baseline in pulse rate at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 62
beats per minute (bpm) | 0.59 (9.706)

8. Primary Outcome: Change From Baseline in Pulse Rate at Week 52
Description: Change from baseline in pulse rate at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 53
bpm | 2.62 (18.441)

9. Primary Outcome: Change From Baseline in Body Weight at Week 24
Description: Change from baseline in body weight at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 64
kilograms (kg) | 0.25 (6.353)

10. Primary Outcome: Change From Baseline in Body Weight at Week 52
Description: Change from baseline in body weight at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 56
kg | -0.16 (8.200)

11. Primary Outcome: Number of Participants With Treatment-emergent Marked Laboratory Abnormalities (MLAs) up to 30 Days After Study Treatment Discontinuation
Description: Number of participants with treatment-emergent MLAs (Hemoglobin [grams/Liter{L}], Hematocrit [L/L], Leukocytes [10^9cells/L], Lymphocytes [10^9cells/L], Alanine Aminotransferase [Units/L {U/L}], Aspartate Aminotransferase [U/L], Bilirubin [micromoles/L {mcmol/L}], Alkaline Phosphatase [U/L], Creatinine [mcmol/L], Urea Nitrogen [mmol/L], Urate [mcmol/L], Potassium [mmol/L], Sodium [mmol/L], Magnesium [mmol/L], Calcium [mmol/L] were reported. Abnormalities that occurred after study treatment start and up to 30 days after study treatment discontinuation, that were not present at baseline, were treatment-emergent. Here, > signifies greater than; < signifies less than; ULN signifies upper limit of normal; and L=Low, H=High, LL=low/low, HH=high/high, LLL=lower/worse than LL, HHH=higher/worse than HH.
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 0.4 to 126 weeks)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 85
Participants
  Hemoglobin:LL<100 | 10
  Hematocrit: LL(<0.28-females;<0.32-males) | 5
  Leukocytes: HH (>20.0) | 1
  Lymphocytes: LLL (<0.5) | 1
  Lymphocytes: LL (<0.8) | 10
  Alanine Aminotransferase: HH (>3 ULN) | 1
  Aspartate Aminotransferase: HH (>3 ULN) | 1
  Alkaline Phosphatase: HH (>2.5 ULN) | 1
  Bilirubin: HH (>2 ULN) | 1
  Bilirubin: HHH (>5 ULN) | 1
  Creatinine: HH (>1.5 ULN) | 2
  Urea Nitrogen: HH (>2.5 ULN) | 3
  Urate: HH (>590) | 15
  Urate: HHH (>720) | 3
  Sodium: LLL (<130) | 3
  Potassium: LLL (<3.0) | 1
  Potassium: LL (<3.2) | 5
  Potassium: HH (>5.5) | 5
  Magnesium: HHH (>1.23) | 1
  Calcium: LLL (<1.75) | 1
  Calcium: LL (<2.0) | 2

12. Primary Outcome: Change From Baseline in Hemoglobin at Week 24
Description: Change from baseline in hemoglobin at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 59
grams per liter (g/L) | -4.13 (11.324)

13. Primary Outcome: Change From Baseline in Hemoglobin at Week 52
Description: Change from baseline in hemoglobin at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 51
grams per litre (g/L) | -1.10 (13.241)

14. Primary Outcome: Change From Baseline in Leukocytes and Platelets at Week 24
Description: Change from baseline in leukocytes and platelets at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 59
10^9 cells/L
  Leukocytes | -0.078 (1.6871)
  Platelets | 1.39 (36.102)

15. Primary Outcome: Change From Baseline in Leukocytes and Platelets at Week 52
Description: Change from baseline in leukocytes and platelets at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 51
10^9 cells/L
  Leukocytes | -0.503 (1.5090)
  Platelets | -9.02 (37.285)

16. Primary Outcome: Change From Baseline in Alanine Aminotransferase and Aspartate Aminotransferase at Week 24
Description: Change from baseline in alanine aminotransferase and aspartate aminotransferase at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: The safety analysis set included all participants who received at least 1 dose of macitentan 10 mg. Here, "N" (number of participants analyzed) specifies number of participants evaluable for this outcome measure; "n" specifies those participants who were analyzed for specific category.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 59
units per liter (U/L)
  Alanine Aminotransferase | -0.49 (7.590)
  Aspartate Aminotransferase: number analyzed (Participants) | 58
  Aspartate Aminotransferase | -0.2 (7.76)

17. Primary Outcome: Change From Baseline in Alanine Aminotransferase and Aspartate Aminotransferase at Week 52
Description: Change from baseline in alanine aminotransferase and aspartate aminotransferase at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 51
U/L
  Alanine Aminotransferase | 0.10 (7.529)
  Aspartate Aminotransferase | 1.2 (6.52)

18. Primary Outcome: Change From Baseline in Bilirubin at Week 24
Description: Change from baseline in bilirubin at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: micromoles per liter (mcmol/L)
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 58
micromoles per liter (mcmol/L) | -0.0970 (4.20548)

19. Primary Outcome: Change From Baseline in Bilirubin at Week 52
Description: Change from baseline in bilirubin at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 49
mcmol/L | 0.2041 (4.65018)

20. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 24
Description: Change from baseline in eGFR rate at Week 24 was reported.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliters/minute/1.73 meter square
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 59
milliliters/minute/1.73 meter square | -4.05 (11.766)

21. Primary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) at Week 52
Description: Change from baseline in eGFR rate at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliters/minute/1.73 meter square
Arm/Group | Macitentan 10 mg
Number analyzed (Participants) | 51
milliliters/minute/1.73 meter square | -1.80 (13.510)

ADVERSE EVENTS:
Time Frame: Up to 30 days after study treatment discontinuation (treatment exposure ranged from 0.4 to 126 weeks)
Description: The safety analysis set included all participants who received at least 1 dose of macitentan 10 milligrams (mg).
Arm/Group | Macitentan 10 mg
All-Cause Mortality (participants affected / at risk) | 11/91
Serious Adverse Events (participants affected / at risk) | 49/91
Other Adverse Events (participants affected / at risk) | 45/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=91)
Anaemia (Blood and lymphatic system disorders) | 2
Acute Left Ventricular Failure (Cardiac disorders) | 1
Angina Pectoris (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 2
Atrioventricular Block Complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure Acute (Cardiac disorders) | 1
Cardiac Failure Chronic (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 6
Left Ventricular Failure (Cardiac disorders) | 3
Right Ventricular Failure (Cardiac disorders) | 5
Sinus Node Dysfunction (Cardiac disorders) | 1
Retinal Vein Thrombosis (Eye disorders) | 1
Abdominal Incarcerated Hernia (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
Death (General disorders) | 1
No Adverse Event (General disorders) | 1
Non-Cardiac Chest Pain (General disorders) | 1
Ulcer Haemorrhage (General disorders) | 1
Cholecystitis Acute (Hepatobiliary disorders) | 2
Cellulitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 1
Covid-19 Pneumonia (Infections and infestations) | 3
Herpes Zoster (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Pneumonia Viral (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Limb Injury (Injury, poisoning and procedural complications) | 1
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1
Blood Potassium Increased (Investigations) | 1
International Normalised Ratio Increased (Investigations) | 1
Sars-Cov-2 Test Positive (Investigations) | 1
Fluid Retention (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Neoplasm of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular Accident (Nervous system disorders) | 2
Ischaemic Stroke (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 5
Renal Impairment (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac Pacemaker Replacement (Surgical and medical procedures) | 1
Cholecystectomy (Surgical and medical procedures) | 1
Small Intestinal Resection (Surgical and medical procedures) | 1
Thyroidectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 10 mg (N=91)
Anaemia (Blood and lymphatic system disorders) | 6
Right Ventricular Failure (Cardiac disorders) | 6
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Oedema Peripheral (General disorders) | 7
Upper Respiratory Tract Infection (Infections and infestations) | 5
Urinary Tract Infection (Infections and infestations) | 9
Haemoglobin Decreased (Investigations) | 5
Weight Increased (Investigations) | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Hypotension (Vascular disorders) | 5

LIMITATIONS AND CAVEATS:
Limited number of efficacy parameters were assessed in an exploratory manner. Study was stopped prematurely as main double-blind study did not meet the primary efficacy outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 30 days before submission for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2020-11-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT03714815/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/15/NCT03714815/SAP_001.pdf